CLINICAL TRIAL: NCT03848039
Title: A Randomised, Double-Blind, Placebo-Controlled, Phase III Study to Investigate the Efficacy of Presurgical 9-valent HPV Vaccination in Women Treated With LEEP for CIN 2+ and Initially Invasive Cervical Cancer.
Brief Title: Impact on Disease Relapse of HPV Vaccination in Women Treated With LEEP for Cervical Intraepithelial Neoplasia. HOPE9
Acronym: HOPE9
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alessandro Ghelardi (Other)
Responsible Party: Sponsor-Investigator, Alessandro Ghelardi, Principal Investigator, Department of Obstetrics and Gynaecology Azienda USL Toscana Nord Ovest, Presidio Ospedaliero delle Apuane (MS)- Italy, Azienda USL Toscana Nord Ovest
Organization: Azienda USL Toscana Nord Ovest (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HOPE9 STUDY; 2018-003507-19 (EudraCT Number)
Record Dates: First submitted 2019-02-19; First posted 2019-02-20 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Cervical Intraepithelial Neoplasia
Keywords: Cervical Cancer; cervical intraepithelial neoplasia; Papillomavirus Vaccines
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gardasil-9 (Experimental): Intramuscular Gardasil-9 vaccination at 0, 2 and 6 months.
  Interventions: Biological: Gardasil-9
- Placebo (Placebo Comparator): Placebo injection at 0, 2 and 6 months
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Gardasil-9 — administration by intramuscular injection of the 9-valent HPV vaccine according to a 3-dose vaccination schedule (0, 2, 6 months).
  Other Names: 9-valent HPV vaccine; Vaccine against HPV-6, 11, 16, 18, 31, 33, 45, 52, 58
  Arms: Gardasil-9
Drug: Placebo — administration by intramuscular injection of the placebo according to vaccination schedule of the 9-valent HPV vaccine (0, 2, 6 months)
  Other Names: Sterile Water for Injection Ph. Eur.
  Arms: Placebo

SUMMARY:
This study evaluates the impact on disease relapse of presurgical 9-valent HPV vaccination versus placebo vaccination in women treated with LEEP (loop electrosurgical excision procedure) for CIN2+ (high grade cervical intraepithelial neoplasia) and initially invasive cervical cancer.

DETAILED DESCRIPTION:
Rationale:

In 2006 HPV vaccination was licensed for primary prevention programs worldwide. Only a few years after, several studies have raised new scenarios about HPV related diseases with strong implications on clinical management in adult women. Some findings from retrospective data have shown a significant effect of HPV vaccine on women and men treated for HPV pathologies. Although vaccination is not effective in patients with prevalent HPV infection, some studies have suggested that HPV vaccine could influence the incidence of the disease relapse after a surgical treatment. Reduction in disease recurrence after surgical treatment in vaccinated patients comes from gastroenterological, gynecological and dermatological evidences concerning both benign lesions (warts) and precancerous lesions.

If vaccination reduces recurrence rates by 80%, according to our previous pilot study data, peri-surgical HPV vaccination will be a strong effective clinical intervention, very likely to be introduced into standard high grade cervical intraepithelial neoplasia management.

Objective:

The primary objective of the current study is to assess the efficacy of 9-valent HPV vaccination in preventing recurrence of CIN2+ in participants treated for high-grade CIN.

Study population: participants treated for CIN2+ with LEEP technique. Study design: A multicenter, randomised, double-blind clinical trial in 9 hospitals in Italy.

Intervention: Participants will be randomized in a 1:1 ratio to receive presurgical 9-valent HPV vaccination (Gardasil-9 ®) or placebo at months 0 (at pre-surgical enrollment time), at 2 months (the same day of surgical treatment) and 6 moths (during the first follow-up visit after surgery). The randomization list will be generated before the start of the study.

Main study parameters/endpoints:

Primary end point will be the cumulative recurrence of CIN2+ after conization, as assessed by biopsies taken of suspect lesions, histologically confirmed for high grade cervical intraepithelial neoplasia recurrence.

Secondary outcome measures are cumulative incidence/persistence of HPV infection after the surgical treatment, causative HPV type in recurrent CIN lesions, as assessed by HPV test and PCR (polymerase chain reaction).

The total sample size is estimated to be 1220 patients based on an expected recurrence rate of less than 6% within 5 years. Statistical analysis will be based on the intention-to-treat protocol. Both primary and secondary endpoints will be analyzed by descriptive statistics and the chi-square test with a 0,05 two-sided significance level.

Follow-up schedule (FUP) will be the same in both arms, with a FUP evaluation every 6 months in the first year followed by an annual evaluation for a total of 5 years. FUP visit will include HPV test, Pap-test and colposcopy. HPV test will be collected in order to evaluate the HPV infection clearance rate in both arms. HPV test will be part of all the follow-up visits allowing to study the natural history of HPV infection after the surgical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 and ecog performance status ≤ 1
2. Patients with a diagnosis of high-grade cervical intraepithelial neoplasia or initially invasive cervical cancer (histological results ≥ CIN2 + and ≤ Ia1 according to the FIGO staging of cervical cancer)
3. No fever at the time of vaccination
4. No previous HPV vaccination
5. Ability to understand and write Italian
6. Signed informed and privacy consent

Exclusion Criteria:

1. Patients enrolled in other clinical studies
2. History of allergic reaction or serious adverse events to previous vaccinations
3. Positive pregnancy test at the time of vaccination
4. Patient in treatment with immunosuppressive therapy
5. Subjects who received immunoglobulins or blood products in 3 months prior to vaccination.
6. Thrombocytopenia or any other clotting disorder that may lead to bleeding as a result of intramuscular administration
7. Clinical criteria contraindicating the surgical act of conization
8. ECOG performance status ≥2

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220 (Estimated)
Dates: Start 2020-12 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2028-05 (Estimated)

PRIMARY OUTCOMES:
evaluation of disease recurrence reduction (cervical intraepithelial neoplasia up to microinvasive cancer of the cervix) | 5 years after surgical treatment
  evaluation of disease recurrence reduction (cervical intraepithelial neoplasia up to microinvasive cancer of the cervix) by comparing the number of recurrences in the two arms of the study

SECONDARY OUTCOMES:
impact of the vaccine on prevalent post-surgery infections | 5 years after surgical treatment
  Analysis of the impact of the vaccine on prevalent post-surgery infections by comparing the prevalence of persistent HPV infections (duration greater than 12 months after surgery) in the two arms.
impact of the vaccine in the post-surgical surveillance times, comparison of viral wash-out times (negativity of the HPV test), times of negativization of the pap test and of the colposcopic picture in the post-operative period | 5 years after surgical treatment
  Analysis of the impact of the vaccine in the post-surgical surveillance times, comparison of the viral wash-out times (negativity of the HPV test), times of negativization of the pap test and of the colposcopic picture in the post-operative period: comparison of the times of negativization overexposed in the two arms.

CONTACTS AND LOCATIONS:
Overall Officials: Alessandro Ghelardi, MD, Principal Investigator — Az. USL Toscana Nord Ovest

IPD SHARING:
Plan to Share IPD: No